CLINICAL TRIAL: NCT05832775
Title: A First-in-human, Double-blind, Placebo-controlled, Multicentre, Cross-over, Phase I Study to Assess Safety and Tolerability of Repeat Oral Administrations of MRx0029 OR MRx0005 in Adult Participants With Idiopathic Parkinson's Disease
Brief Title: Study to Assess the Safety of MRx0029 or MRx0005 Compared to Placebo, in People With Parkinson's
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor insolvency
Sponsor: 4D pharma plc (Industry)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry); ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INNOVATE-LBP 1.0
Record Dates: First submitted 2022-03-08; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Microbiome
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MRx0029 Treatment Sequence 1 (Experimental): Patients will receive MRx0029 in the first treatment period and then placebo in the second treatment period
  Interventions: Biological: MRx0029
- MRx0029 Treatment Sequence 2 (Experimental): Patients will receive placebo in the first treatment period and then MRx0029 in the second treatment period
  Interventions: Biological: MRx0029
- MRx0005 Treatment Sequence 1 (Experimental): Patients will receive MRx0005 in the first treatment period and then placebo in the second treatment period
  Interventions: Biological: MRx0005
- MRx0005 Treatment Sequence 2 (Experimental): Patients will receive placebo in the first treatment period and then MRx0005 in the second treatment period
  Interventions: Biological: MRx0005

INTERVENTIONS:
Biological: MRx0029 — Megasphaera massiliensis MRx0029 (Treatment A) and Placebo
  Arms: MRx0029 Treatment Sequence 1; MRx0029 Treatment Sequence 2
Biological: MRx0005 — Parabacteroides distasonis MRx0005 (Treatment B) and Placebo
  Arms: MRx0005 Treatment Sequence 1; MRx0005 Treatment Sequence 2

SUMMARY:
This is a first-in-human study to evaluate the safety and tolerability of repeat oral administrations of MRx0029 (20 participants) or MRx0005 (20 participants) in participants diagnosed with idiopathic PD. Participants who are successfully screened will be randomized to 1 of 2 treatment sequences (TS) within their cohort (10 participants per sequence). Each treatment period will be separated by a washout period of 4 to 6 weeks.

Cohort A Treatment Sequence 1: MRx0029 (1 capsule bid) for 4 weeks; 4-to 6-week washout period; placebo (1 capsule bid) for 4 weeks.

Cohort A Treatment Sequence 2: Placebo (1 capsule bid) for 4 weeks; 4-to 6-week washout period; MRx0029 (1 capsule bid) for 4 weeks.

Cohort B Treatment Sequence 1 MRx0005 (1 capsule bid) for 4 weeks; 4- to 6-week washout period; placebo (1 capsule bid) for 4 weeks.

Cohort B Treatment Sequence 2: Placebo (1 capsule bid) for 4 weeks; 4-to 6-week washout period; MRx0005 (1 capsule bid) for 4 weeks

Cohort A will be randomized first and when all participants have been randomized to Cohort A, Cohort B enrollment will begin.

DETAILED DESCRIPTION:
There will be a total of 10 visits which will include a screening visit, 8 treatment period visits, and a Follow-up Visit. Three telephone calls will be made during the study to assess the participant's health status and confirm eDiary compliance. Participants will be screened for eligibility between Day -28 to Day -2 (Visit 1, screening). Informed consent will be obtained before performing any study-related procedures.

Following randomization, participants will be provided with enough study medication to administer at home for 4 weeks (+/-2 days). The participants will discontinue treatment for 4 to 6 weeks. The participants will return to the site for the second period of study treatment and will again be provided with enough study medication to administer at home for 4 weeks (+/-2 days).

Frequency of the AEs monitored throughout the study, and changes in laboratory values, vital signs, ECGs, and physical examinations will be assessed at the beginning and at the end of each treatment period.

Gut permeability will be assessed with administration of a sugar solution and subsequent 24 hour urine collection.

During the study, participants will report their daily bowel habits, including stool consistency, with the use of an electronic diary (the Bristol Stool Chart diary). The participants will also provide a stool sample on Day 1 and Day 29 of each treatment period and at the Follow-up Visit.

PD symptoms will be assessed with the use of MDS-UPDRS and MDS-NMS to confirm that MRx0005 and MRx0029 do not adversely impact a participant's Parkinson's symptoms.

Participants will report their dietary habits by filling out a Food Frequency Questionnaire at the clinic visits beginning (Day 1) and at the end of each treatment period, and at the Follow-up Visit.

For the participants who are on stable immediate release formulations of levodopa, PK of levodopa will be assessed at the beginning (Day 1, prior to the first IMP dosing) and at the end (Day 29) of each treatment period.

Fecal microbiome, as well as plasma/serum, fecal and urine biomarkers will be assessed, on Day 1 prior to the start of each treatment (baseline) period and at the end of each treatment period (Day 29), and at the Follow-up Visit.

Participants will undergo a 4- to 6-week washout between treatment periods. Approximately 4 to 6 weeks after their second EOT visit, the participants will attend the clinic for their Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD according to the UKPDS-BBCDC
2. Able to understand and willing to provide informed consent and able to comply with the study procedures and restrictions.
3. Male or female participants age ≥ 40 or ≤ 85 years of age.
4. BMI ≥ 18.0 to ≤ 35.0 kg/m2, inclusive, where BMI (kg/m2) is calculated by body weight (kg)/height2 (m2).
5. Hoehn & Yahr (H&Y) Stage I to II (if on levodopa the participant should be classed as Stage I to II in an 'ON' period)
6. A documented diagnosis of PD
7. If presently being medically treated for PD, they should be on a stable dose unchanged within the 30 days prior to screening and not be expected to require any adjustments or start any new PD medication for the duration of their participation in the study.
8. No clinically relevant abnormal medical history, or abnormal findings on physical examination, vital signs, ECG, or laboratory tests
9. Has been fully vaccinated with an approved Covid-19 vaccine
10. Male and female participants are eligible to enter provided they follow the contraception criteria for the study.

Exclusion Criteria:

1. Participants with significant motor fluctuations
2. Parkinson syndromes
3. Known carriers of familial PD genes
4. History and/or current presence of clinically significant CNS disease other than PD.
5. Montreal Cognitive Assessment (MoCA) <24
6. No history of spontaneous constipation since diagnosis
7. Participants who are <70% compliant to completing their e-daily assessed at Treatment Period 1, Day 1.
8. Are non-compliant with prescribed PD medication
9. Comorbidities that have not been optimally controlled for the last 3 months prior to screening.
10. Participants with known Type 1 or Type 2 diabetes mellitus or a HbAlc result. indicative of diabetes/pre-diabetes.
11. Have an active or recent malignant disease or any concomitant end-stage organ disease.
12. Participants with known GI fistula, feeding tubes, or inflammatory bowel disease.
13. Participants who had recent abdominal surgery (6 months before the screening visit).
14. Participants with GI disease resulting in an inability to take oral medication, malabsorption syndrome, prior surgical procedures affecting absorption, uncontrolled GI disease
15. Participants with conditions that may increase the risk of generalized peritonitis
16. Dysphagia to the extent it would affect the participant's ability to swallow the IMP during their participation
17. Anything which in the opinion of the investigator prevents the participant being able to give urine or stool samples.
18. Positive serology for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV), or human immunodeficiency virus antibodies (anti HIV) 1/2 at screening.
19. Previous history or current active tuberculosis (TB), or taking medication for the treatment of TB.
20. Participant has severe or moderate renal impairment (defined as creatinine clearance <60 mL/min) estimated using Cockcroft-Gault Equation.
21. Participants taking anti-cholinergic medication or amantadine.
22. Participants with congenital, acquired or drug-related immunodeficiency.
23. Participants who use systemic corticosteroids or systemic immunosuppressants for any reason within 30 days prior to screening.
24. Participants taking ad hoc anti-inflammatory medication within 30 days of screening are excluded.
25. Participants taking dopamine antagonists, such as the neuroleptics or metoclopramide are excluded.
26. Participants who are allergic to the following antibiotics: amoxicillin/clavulanic acid, ampicillin, chloramphenicol, clarithromycin, clindamycin, imipenem, or metronidazole.
27. Participants who have completed a course of systemic antibiotics in the 30 days prior to screening.
28. Participants using prebiotic and probiotic supplements
29. Donation or loss of 500 mL blood during the 3 months before screening.
30. Current or history of alcohol or drug abuse or other dependence (except nicotine dependence) within the last 2 years prior to IMP administration.
31. Positive urine drug screen (if not due to concomitant medication) or alcohol breath test.
32. Receipt of a positive COVID-19 test result
33. Participant is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or study drug(s), or participant receiving other investigational agent(s).
34. Received a live vaccine within 4 weeks prior to enrolling in this trial or plan for any such vaccination during the trial or within 4 months after study drug administration. Administration of inactivated vaccines (for example, inactivated influenza vaccines is allowed.).
35. Legal incapacity or limited legal capacity.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Baseline to Follow-up Visit (up to 24 weeks)
  Number of TEAEs after 4-weeks of treatment with MRx0029 vs 4-weeks of placebo in participants with idiopathic PD
Incidence of treatment-emergent adverse events (TEAEs) | Baseline to Follow-up Visit (up to 24 weeks)
  Number of TEAEs after 4 weeks of treatment with MRx0005 vs 4-weeks of placebo in participants with idiopathic PD
Incidence of Serious Adverse Events (SAEs) | Baseline to Follow-up Visit (up to 24 weeks)
  Number of SAEs after 4 weeks of treatment with MRx0029 vs 4-weeks of placebo in participants with idiopathic PD
Incidence of Serious Adverse Events (SAEs) | Baseline to Follow-up Visit (up to 24 weeks)
  Number of SAEs after 4 weeks of treatment with MRx0005 vs 4-weeks of placebo in participants with idiopathic PD

IPD SHARING:
Plan to Share IPD: No